CLINICAL TRIAL: NCT00159562
Title: Effects of Psycho-education of Patients With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Norwegian Council for Mental Health (Other); Norwegian Foundation for Health and Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EW-2005
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2015-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Psycho-education
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group education (Experimental): Bipolar 1 and 2 patients in a stable euthymic phase will receive group education in 10 weekly sessions and then a session every third month for two years. Symptoms, admittances to hospital and function will be followed for two years.
  Interventions: Behavioral: Group education
- individual education (Active Comparator): Bipolar 1 and 2 patients in a stable euthymic phase will receive three individual sessions of education.
  Interventions: Behavioral: individual education

INTERVENTIONS:
Behavioral: individual education — individual sessions of psycho-education
  Arms: individual education
Behavioral: Group education — group psycho-education in 10 weekly sessions and then a session every third month for two years
  Arms: group education

SUMMARY:
The purpose for this study is to determine whether psycho-education in groups is more effective than individual psycho-education for patients with bipolar disorder.

DETAILED DESCRIPTION:
The main aim of the study is to compare the effects of psycho-education in groups with short individual psycho-education.

It is a randomized controlled trial including Bipolar 1 and 2 patients in a stable euthymic phase. 42 or 43 patients will receive group education in 10 weekly sessions and then a session every third month for two years. 42 or 43 patients will receive three individual sessions of education. Symptoms, admittances to hospital and function will be followed for two years.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar Disorder 1 or 2 Euthymic

Exclusion Criteria:

* Active depression or mania/hypomania

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2005-09; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Score on depression and mania rating scales | 12 months
Admissions to hospital | 24 months
Working activity | 24 months

SECONDARY OUTCOMES:
Symptoms, function, use and change in medication, need for | 24 months
consultations | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Morken, PhD MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Østmarka Psychiatric Department, St Olavs Hospital, University Hospital of Trondheim, Trondheim, Norway

REFERENCES:
- [Result] Kallestad H, Wullum E, Scott J, Stiles TC, Morken G. The long-term outcomes of an effectiveness trial of group versus individual psychoeducation for bipolar disorders. J Affect Disord. 2016 Sep 15;202:32-8. doi: 10.1016/j.jad.2016.05.043. Epub 2016 May 24. PMID 27253214